CLINICAL TRIAL: NCT00734565
Title: A Phase I, Single-arm, Single-center Study to Investigate Safety and Reactogenicity of Monovalent Conjugated Vaccine Against Haemophilus Influenzae Type b in Healthy Children Aged 16 - 20 Months and Infants Aged 2 - 4 Months
Brief Title: Safety and Reactogenicity of a Monovalent Conjugated Vaccine Against Haemophilus Influenzae Type b
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: M37P1
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Haemophilus Influenzae Type b
Keywords: vaccine; prevention; haemophilus influenzae type b; children
MeSH Terms: conditions — Haemophilus Infections

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Haemophilus influenzae type b

INTERVENTIONS:
Biological: Haemophilus influenzae type b — 1 dose monovalent conjugated vaccine against Haemophilus influenzae type b in children aged 16 - 20 months and infants aged 2 - 4 months

SUMMARY:
This study will investigate safety and reactogenicity of a monovalent conjugated vaccine against Haemophilus influenzae type b in healthy children

ELIGIBILITY:
Inclusion Criteria:

* Infants of either sex, aged 16 - 20 months / 2 - 4 months
* in good health as determined by: medical history physical examination clinical judgment of the investigator;
* available for all visits scheduled in the study and able to comply with all study regulations;
* written informed consent obtained, from at least one parent or legal guardian

Exclusion Criteria:

* parent or legal guardian is unwilling or unable to give written informed consent to participate in study;
* infants who presented a previous disease potentially related to Haemophilus influenzae type b;
* infants who had household contact and/or intimate exposure in the previous 30 days to an individual with ascertained Haemophilus influenzae type b disease;
* infants who have received any other Haemophilus influenzae type b immunization dose before (for 16-20 months old children who have received a booster vaccination already);
* premature (before 37th week of gestation) or birth weight less than 2500 g;
* history of anaphylactic shock, asthma, urticaria or other allergic reaction after previous vaccinations or hypersensitivity to any vaccine component;
* fever ≥38.0 °C (axillary body temperature) and/or significant acute or chronic infection requiring systemic antibiotic or antiviral therapy within the past 7 days before enrollment;
* subjects with any serious chronic disease such as cardiac, neurological, metabolic, hematologic, or neoplastic disease;
* known/suspected immunodeficiency, or autoimmune disease, or any immunologic disorder;
* subjects with any neurological disorder, e.g., epilepsy or history of seizure disorder;
* subjects with a clinically significant genetic anomaly;
* treatment with corticosteroids or other immunosuppressive drugs;
* treatment with parenteral immunoglobulin preparation, blood products, and/or plasma derivatives (or: within the past 3 months - applicable for children 16 - 20 months);
* any vaccination administered within 2 weeks (14 days) before enrollment;
* participation in any other investigational trial simultaneously;
* planned surgery during the study period;
* any condition, which, in the opinion of the investigator, might interfere with the evaluation of the study objective

Ages: 2 Months to 20 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2008-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Rates of local and systemic reactions, adverse events (AEs), and serious adverse events (SAEs) after first vaccination dose will be evaluated. | 30 days

SECONDARY OUTCOMES:
Rates of local and systemic reactions, adverse events (AEs), and serious adverse events (SAEs) after second vaccination dose will be evaluated. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- Vaccination site, Shijiazhuang, China